CLINICAL TRIAL: NCT00950755
Title: Phase II Study of Iodine 131 Anti B1 Antibody for 1st or 2nd Relapsed Indolent B-Cell Lymphomas or B-Cell Lymphomas That Have Transformed to a More Aggressive Histology
Brief Title: Study of Iodine 131 Anti B1 Antibody for 1st or 2nd Relapsed Indolent B-Cell Lymphomas or B-Cell Lymphomas That Have Transformed to a More Aggressive Histology
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104505
Record Dates: First submitted 2009-07-30; First posted 2009-08-03 (Estimated); Results first posted 2012-08-29 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-11

CONDITIONS: Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — tositumomab I-131

ARMS (1):
- Tositumomab and Iodine I 131 Tositumomab (anti-B1 antibody) (Experimental): In the first phase (dosimetric dose) patients will receive an infusion of unlabeled Anti B1 Antibody (450 mg) followed by an infusion of Anti B1 Antibody (35 mg) which has been trace-labeled with 5 mCi of Iodine 131. Whole body gamma camera scans will be obtained following the dosimetric dose. Using the dosimetric data, a patient-specific dose of Iodine 131 Anti B1 Antibody to deliver the desired total body dose of radiotherapy will be calculated. In the second phase, (radioimmunotherapeutic dose), patients will receive an infusion of unlabeled Anti B1 Antibody (450 mg) followed by an infusion of 35 mg Anti B1 Antibody labeled with the patient-specific dose of Iodine 131 to deliver a whole body dose of 75 cGy. Patients will be treated with saturated solution potassium iodide, Lugol's solution, or potassium iodide tablets starting at least 24 hours prior to the first infusion and continuing for 14 days following the last infusion of Iodine 131 Anti B1 Antibody.
  Interventions: Biological: tositumomab and Iodine I 131 tositumomab (anti-B1 antibody)

INTERVENTIONS:
Biological: tositumomab and Iodine I 131 tositumomab (anti-B1 antibody) — For the treatment of 1st or 2nd relapsed indolent B cell lymphomas or B cell lymphomas that have transformed to a more aggressive histology

SUMMARY:
This is a single-arm, open-label study of Iodine 131 Anti B1 Antibody for the treatment of 1st or 2nd relapsed indolent B cell lymphomas or B cell lymphomas that have transformed to a more aggressive histology. The primary endpoint of the study is to determine the response rate. Secondary endpoints of the study is to determine the duration of response, time to progression, time-to-treatment failure, safety, and survival.

Forty patients will receive therapy on this study at the 2 clinical sites. Patients will undergo 2 phases of the study. In the first phase, termed the "dosimetric dose", patients will receive an infusion of unlabeled Anti B1 Antibody (450 mg) over 70 minutes (including a 10 minute flush) immediately followed by a 30 minute infusion (including a 10 minute flush) of Anti B1 Antibody (35 mg) which has been trace-labeled with 5 mCi of Iodine 131. Whole body gamma camera scans will be obtained on 1) Day 0; 2) Day 2, 3, or 4; and 3) Day 6 or 7 following the dosimetric dose. Using the dosimetric data from the 3 imaging timepoints, a patient-specific dose of Iodine 131 Anti B1 Antibody to deliver the desired total body dose of radiotherapy will be calculated. In the second phase, termed the "radioimmunotherapeutic dose", patients will receive a 70 minute infusion (including a 10 minute flush) of unlabeled Anti B1 Antibody (450 mg) immediately followed by a 30 minute infusion (including a 10 minute flush) of 35 mg Anti B1 Antibody labeled with the patient-specific dose of Iodine 131 to deliver a whole body dose of 75 cGy to patients with no hematologic risk factors. Patients who have platelet counts of 100,001-149,999 cells/mm3 will receive 65 cGy and patients who are obese will be dosed based upon 137% of their lean body mass (see Appendix A). Patients will be treated with either saturated solution potassium iodide (SSKI), Lugol's solution, or potassium iodide tablets starting at least 24 hours prior to the first infusion of the Iodine 131 Anti B1 Antibody and continuing for 14 days following the last infusion of Iodine 131 Anti B1 Antibody (i.e., therapeutic dose).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically-confirmed diagnosis of B-cell CLL/PLL/SLL; lymphoplasmacytic - immunocytoma; follicle center, follicular, grade I; or follicle center, follicular, grade II NHLs or one of these B-cell lymphomas which has transformed to a more aggressive histology (37).
* Patients must have evidence that their tumor tissue expresses the CD20 antigen. Immunoperoxidase stains of paraffin-embedded tissue showing positive reactivity with L26 antibody or immunoperoxidase stains of frozen tissue showing positive reactivity with Anti B1 Antibody (>50% of tumor cells are positive) or evidence of CD20 positivity by flow cytometry (>50% of tumor cells are positive) are acceptable evidence of CD20 positivity. Testing of tumor tissue from any time in the course of the patient's disease is acceptable.
* Patients must have received 1 or 2 prior chemotherapy regimens and have progressed following their last regimen. Patients who have received >2 prior chemotherapy regimens are excluded. Prior therapy with radiation, immunosuppressants, or steroids are not counted as chemotherapy regimens.
* Patients must have a performance status of at least 60% on the Karnofsky Scale (see Appendix B) and an anticipated survival of at least 3 months.
* Patients must have an absolute granulocyte count >1,500 x 109/l and a platelet count >100,000 x 109/l within 14 days of study entry. These blood counts must be sustained without support of hematopoietic cytokines or transfusion of blood products.
* Patients must have adequate renal function (defined as serum creatinine <1.5 upper limit of normal) and hepatic function (defined as total bilirubin <1.5 upper limit of normal and hepatic transaminases [AST + ALT] <5 x upper limit of normal) within 14 days of study entry.
* Patients must have bi-dimensionally measurable disease. At least one lesion must be >/=2cm x 2 cm (by CT scan).
* Patients must be at least 18 years of age.
* Patients must give written informed consent and sign an EC-approved informed consent form prior to study entry.

Exclusion Criteria:

* Patients with more than an average of 25% of the intratrabecular marrow space involved by lymphoma in bone marrow biopsy specimens as assessed microscopically within 42 days of study entry. Bilateral posterior iliac crest core biopsies are required if the percentage of intratrabecular space involved exceeds 10% on a unilateral biopsy. The mean of bilateral biopsies must be no more than 25%. The procedure for bilateral bone marrow biopsy analysis of marrow involvement is included in Appendix C.
* Patients who have received cytotoxic chemotherapy, radiation therapy, or cytokine treatment within 4 weeks prior to study entry (6 weeks for nitrosourea compounds) or who exhibit persistent clinical evidence of toxicity. The use of systemic steroids must be discontinued one week prior to study entry.
* Patients with prior hematopoietic stem cell transplant following high-dose chemotherapy or chemo/radiotherapy.
* Patients with active obstructive hydronephrosis.
* Patients with evidence of active infection requiring IV antibiotics at the time of study entry.
* Patients with New York Heart Association class III or IV heart disease (see Appendix D) or other serious illness that would preclude evaluation.
* Patients with prior malignancy other than lymphoma, except for adequately-treated skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for 5 years. Patients who have been disease-free of another cancer for greater than 5 years must be carefully assessed at the time of study entry to rule out recurrent disease.
* Patients with known HIV infection.
* Patients with known brain or leptomeningeal metastases.
* Patients who are pregnant or breast-feeding. Patients of child-bearing potential must undergo a serum pregnancy test within 7 days prior to study entry and radiolabeled antibody is not to be administered until a negative result is obtained. Males and females must agree to use effective contraception for 6 months following treatment.
* Patients with previous allergic reactions to iodine. This does not include reacting to IV iodine-containing contrast materials.
* Patients who were previously given any monoclonal or polyclonal antibodies of any non-human species for either diagnostic or therapeutic purposes. This includes engineered chimeric and humanized antibodies.
* Patients who previously received radioimmunotherapy.
* Patients with progressive disease within 1 year of irradiation arising in a field that has been previously irradiated with >3500 cGy.
* Patients who are concurrently receiving either approved or non-approved (through another protocol) anti-cancer drugs or biologics.
* Patients who have received more than 2 prior chemotherapy regimens. Prior therapy with radiation, immunosuppressants, or steroids are not counted as chemotherapy regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 1998-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 104505 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104505 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104505 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104505 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 104505 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104505 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104505 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) received radioimmunotherapy of tositumomab (TST) and Iodine I 131 TST in 2 phases (Ph.): Ph. 1, dosimetric dose; Ph. 2, therapeutic dose. Par. were evaluated until disease progression, they died, or they were on study for 2 years. Par. completing 2 years of study could enter a long-term follow-up study (BEX104528; NCT00240578).
Groups:
- TST and Iodine I 131 TST: Participants received a dosimetric dose (DD) consisting of 450 milligrams (mg) of tositumomab (TST) intravenously (IV) followed by 5.0 millicurie (mCi) of Iodine I 131 and 35 mg of TST IV. The therapeutic dose (TD) consisting of 450 mg of TST IV, followed by a participant-specific dose of I 131 (75 centigray [cGy] or 65 cGy) and 35 mg of TST IV, was administered 7-14 days after the DD. Participants who had disease progression or had completed at least 2 years of follow-up after administration of TST/I 131 TST during the TD phase and had signed the informed consent to participate in the Long-Term Follow-Up (LTFU) study (BEX104528) were followed for up to 10 years. Participants did not receive any study medication during the LTFU study.
Period: Dosimetric and Therapeutic Treatment
Arm/Group | TST and Iodine I 131 TST
Started | 41
Completed | 0
Not Completed | 41
Not completed — Lost to Follow-up | 3
Not completed — Received Alternative Therapy | 1
Not completed — Progressive Disease | 27
Not completed — Death | 1
Not completed — Stroke; Difficult to Attend Study Visits | 1
Not completed — Participant Moved; Unable to Follow Up | 1
Not completed — Rolled Over to Study BEX104528 | 6
Not completed — Investigator Discretion | 1
Period: Long-Term Follow-Up
Arm/Group | TST and Iodine I 131 TST
Started | 18 (18 of the 41 participants withdrawing from Study BEX104505 enrolled in the LTFU study.)
Completed | 9
Not Completed | 9
Not completed — Lost to Follow-up | 1
Not completed — Death | 8

BASELINE CHARACTERISTICS:
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.2 (11.4)
Gender [Count of Participants; unit: Participants]
  Female | 21
  Male | 20
Race/Ethnicity, Customized [Number; unit: participants]
  White | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (Par.) With Response as Assessed by the Investigator
Description: Par. with response include those with Complete Response (CR: complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease), Clinical Complete Response (CCR: complete resolution of all disease-related symptoms; residual foci, thought to be residual scar tissue, are present), or Partial Response (PR: >=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions; no new lesions).
Time Frame: Par. were evaluated until death/disease progression or 2 years in Study BEX104505. Par. who completed 2 years in BEX104505 were followed in study BEX104528 for up to 125 months. Data are included from both Study BEX104505 and Study BEX104528.
Population: Intent-to-Treat (ITT) Exposed Population: all participants who were enrolled into the study and received at least one dose of study drug. Only those participants evaluable for response were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 40
participants | 31
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST; Test type: Superiority or Other; percentage of participants = 76, 95% CI 2-sided [62 to 89] — The estimated value represents the percentage of participants with response

2. Primary Outcome: Number of Participants With Confirmed Response as Assessed by the Investigator
Description: Responses had to be confirmed by 2 separate evaluations occurring >=4 weeks apart. Par. with confirmed response include those with Complete Response (CR: complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease), Clinical Complete Response (CCR: complete resolution of all disease-related symptoms; residual foci, thought to be residual scar tissue, are present), or Partial Response (PR: >=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions; no new lesions).
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants evaluable for confirmed response were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 35
participants | 22
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST; Test type: Superiority or Other; percentage of participants = 54, 95% CI 2-sided [38 to 69] — The estimated value represents the percentage of participants with confirmed response

3. Primary Outcome: Number of Participants With Confirmed Complete Response (CR) as Assessed by the Investigator
Description: Responses had to be confirmed by 2 separate evaluations occurring >=4 weeks apart. CR is defined as the complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants evaluable for confirmed response were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 35
participants | 14
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST; Test type: Superiority or Other; percentage of participants = 34, 95% CI 2-sided [20 to 49] — The estimated value represents the percentage of participants with confirmed CR

4. Primary Outcome: Number of Participants With Confirmed Complete Response Plus Clinical Complete Response (CR + CCR) as Assessed by the Investigator
Description: Responses had to be confirmed by 2 separate evaluations occurring >4 weeks apart. CCR is defined as the complete resolution of all disease-related symptoms; residual foci, thought to be residual scar tissue, are present. Generally, an unchanging lesion =<2 centimeters (cm) in diameter by radiographic evaluation or =<1 cm in diameter by physical examination can be considered scar tissue. The extent of disease (EOD) must be unchanged or decreased upon follow-up evaluations. If the EOD was unchanged or if further decreases occurred for >=6 months, the participant was reclassified as having a CR.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants evaluable for CR + CCR were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 35
participants | 17
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST; Test type: Superiority or Other; percentage of participants = 41, 95% CI 2-sided [26 to 57] — The estimated value represents the percentage of participants with confirmed CR + CCR

5. Primary Outcome: Number of Participants With Confirmed Partial Response (PR) as Assessed by the Investigator
Description: Responses had to be confirmed by 2 separate evaluations occurring >=4 weeks apart. Confirmed PR is defined as a >=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions, with no new lesions.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants evaluable for confirmed PR were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 35
participants | 4
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST; Test type: Superiority or Other; percentage of participants = 10, 95% CI 2-sided [1 to 19] — The estimated value represents the percentage of participants with confirmed PR

6. Secondary Outcome: Duration of Response for All Confirmed Responders (CR, CCR, or PR) as Assessed by the Investigator
Description: Responses had to be confirmed by 2 separate evaluations occurring >=4 weeks apart. Duration of response is defined as the time from the first documented response until disease progression. Disease progression is defined as a >=25% increase from the nadir value of the sum of the products of the longest perpendicular diameters of all measurable lesions or the appearance of any new lesion. Individual lesions must be >2 cm in diameter by radiographic evaluation or >1 cm in diameter by physical examination.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants with confirmed response and those who experienced progressive disease were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 13
months | 46.4 [15.2 to NA] — The upper limit of the 95% confidence interval (CI) was not able to be determined (not reached) because there were not enough events to be able to calculate the upper limit of the 95% CI.

7. Secondary Outcome: Time to Progression of Disease or Death as Assessed by the Investigator
Description: Time to progression or progression-free survival is defined as the time from the dosimetric dose to the first documented occurrence of disease progression or death. Disease progression is defined as a >=25% increase from the nadir value of the sum of the products of the longest perpendicular diameters of all measurable lesions or the appearance of any new lesion. New lesions must be greater than 2 x 2 centimeters (cm) in diameter by radiographic evaluation or greater than 1 cm in diameter by physical examination.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants who experienced progression were evaluated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 32
months | 12.6 [6.1 to 29.9]

8. Secondary Outcome: Time to Treatment Failure as Assessed by the Investigator
Description: Time to treatment failure is defined as the length of time from the date of enrollment to the first incidence of treatment withdrawal, study removal, progression, and/or alternative therapy for the participant's lymphoma, or death.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants who experienced treatment failure were evaluated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 33
months | 9.5 [6.0 to 26.9]

9. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the treatment start date to the date of death from any cause.
Time Frame: as for outcome 1
Population: Only those participants who died during the study and during the follow-up period were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 26
months | 74.5 [34.9 to 121.5]

10. Secondary Outcome: Number of Participants With the Indicated Adverse Events (AE) Possibly or Probably Related to Study Drug and Experienced by at Least 5% of Participants
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The Investigator assessed whether the AE was possibly or probably related to study drug. In addition, all laboratory-derived hematologic toxicities were assumed to be possibly or probably related to study drug.
Time Frame: as for outcome 1
Population: ITT Exposed Population
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 41
participants
  Absolute Neutrophil Count (ANC) <1000 cells/cm^3 | 18
  White Blood Cells (WBC) <2000 cells/cm^3 | 14
  Platelets <50000 cells/cm^3 | 15
  Hemoglobin <8.0 grams/deciliter (g/dL) | 3
  Nausea | 12
  Constipation | 3
  Vomiting | 3
  Diarrhea | 2
  Lethargy | 6
  Headache | 4
  Paraesthesia | 3
  Somnolence | 3
  Thrombocytopenia | 11
  Anemia | 7
  Neutropenia | 2
  Pancytopenia | 2
  Fatigue | 6
  Pyrexia | 6
  Chills | 5
  Pain | 3
  Herpes Zoster | 3
  Lower Respiratory Tract Infection | 3
  Pneumonia | 3
  Upper Respiratory Tract Infection | 3
  Neutropenic Sepsis | 2
  Respiratory Tract Infection | 2
  Rhinitis | 2
  Cough | 4
  Oropharyngeal Pain | 4
  Dyspnea | 3
  Sneezing | 2
  Back pain | 2
  Muscle Spasms | 2
  Myalgia | 2
  Rash | 4
  Contusion | 2
  Fall | 2
  Hypothyroidism | 4
  Decreased Appetite | 3
  Myelodysplastic Syndrome | 3
  Orthostatic Hypotension | 2

11. Secondary Outcome: Number of Participants With the Indicated Serious Adverse Events (SAE) Related to Study Drug
Description: An SAE is any event occurring at any dose that results in any of the following: death, a life-threatening adverse drug experience (ADE; at immediate risk of death from the experience as it occurred), inpatient hospitalization/prolongation of existing hospitalization, a persistent/significant disability/incapacity, or a congenital anomaly/birth defect. Medical events that may not result in death, be life-threatening, or require hospitalization may be considered to be a serious ADEs when based upon appropriate medical judgment. Relatedness was based on the Investigator's medical judgement.
Time Frame: as for outcome 1
Population: ITT Exposed Population. All participants who experienced any SAE were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 13
participants
  Anemia | 6
  Thrombocytopenia | 6
  Pancytopenia | 2
  Febrile Neutropenia | 1
  Neutropenia | 1
  Lower Respiratory Tract Infection | 2
  Pneumonia | 2
  Hemophilus Infection | 1
  Herpes Simplex | 1
  Herpes Zoster | 1
  Neutropenic Sepsis | 1
  Respiratory Tract Infection | 1
  Myelodysplastic Syndrome | 3
  Pyrexia | 2
  Hematuria | 1
  Renal Failure Chronic | 1
  Hepatic Failure | 1
  Hypercalcemia | 1
  Radiculitis Brachial | 1

12. Secondary Outcome: Number of Participants With the Indicated Type of Infection
Description: An infection is the colonization of a host organism by a parasite species. Infecting parasites seek to use the host's resources to reproduce, often resulting in disease. Specimen samples of the body fluid are cultured for testing whether the infectious organism is present and grown in the culture media to assess the growth pattern of the organisms present in the specimen. The culture results could be positive or negative. The positive culture results indicate that the tested participant has the infection under investigation, in which case therapeutic treatment with anti-infective is required.
Time Frame: as for outcome 1
Population: ITT Exposed Population
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 41
participants
  Any Infection; n=41 | 21
  No Infection; n=41 | 20
  Meningitis; n=21 | 0
  Pyelonephritis; n=21 | 0
  Sepsis; n=21 | 3
  Pneumonia; n=21 | 1
  Endocarditis/Pericarditis; n=21 | 0
  Peritonitis; n=21 | 0
  Other Infections; n=21 | 20

13. Secondary Outcome: Number of Participants With an Infection for Which Anti-infectives Were Administered
Description: Anti-infectives are capable of acting against infection, by inhibiting the spread of an infectious agent or by killing the infectious agent outright. Anti-infective is a general term that encompasses antibacterials, antibiotics, antifungals, antiprotozoans, and antivirals.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants who had infection during the study and during the follow-up period were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 21
participants
  Anti-infective Administered | 18
  Anti-infective Not Administered | 3

14. Secondary Outcome: Duration of the Indicated Grade 3 or Grade 4 Hematologic Toxicities
Description: Adverse events were graded using the Common Toxicity Criteria from the Cancer Therapy Evaluation Program, Division of Cancer Therapy, National Cancer Institute. Grades: 0 = No adverse event or within normal limits; 1 = Mild adverse event; 2 = Moderate adverse event; 3 = Severe and undesirable adverse event; 4 = Life-threatening or disabling adverse event; 5 = Death related to adverse event.
Time Frame: as for outcome 1
Population: ITT Exposed Population. The "n" in the category titles reflects the number of participants with the indicated Grade 3 or Grade 4 hematologic toxicity.
Measure: Median (Full Range); unit: days
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 41
days
  ANC, n=18 | 16 [5 to 179]
  Hemoglobin, n=3 | 25 [6 to 375]
  Platelets, n=15 | 28 [8 to 261]
  WBC count, n=14 | 23 [8 to 179]

15. Secondary Outcome: Time to Nadir and Time to Recovery to Baseline in Hematologic Laboratory Evaluations
Description: Nadir is defined as the lowest laboratory value recorded following the administration of the study medication. Time to recovery to baseline in hematologic laboratory evaluations is the time required for recovery from nadir values to baseline values.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants with hematologic toxicity were evaluated for time to nadir and time to recovery to baseline. Hematologic toxicity is defined as laboratory values outside the normal range (different for each parameter).
Measure: Median (Full Range); unit: days
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 40
days
  Time to nadir ANC, n=40 | 42.5 [11 to 54]
  Time to nadir hemoglobin, n=40 | 47 [14 to 96]
  Time to nadir platelets, n=40 | 32 [19 to 65]
  Time to nadir WBC count, n=40 | 42.5 [11 to 54]
  Time to recovery to baseline ANC, n=35 | 61 [54 to 85]
  Time to recovery to baseline hemoglobin, n=30 | 61 [54 to 86]
  Time to recovery to baseline platelets, n=35 | 49 [46 to 61]
  Time to recovery to baseline WBC count, n=34 | 85 [57 to 88]

16. Secondary Outcome: Nadir Values for Hematologic Parameters ANC, Platelets, and WBC Count
Description: Nadir is defined as the lowest laboratory value recorded following the administration of study medication. ANC is a measure of the number of neutrophil granulocytes present in the blood. Neutrophils are a type of WBC that fights against infection. Platelets and WBCs are types of blood cells.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants with hematologic toxicity were evaluated. Hematologic toxicity is defined as laboratory values outside the normal range (different for each parameter).
Measure: Median (Full Range); unit: 1000 cells/millimeters cubed (mm^3)
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 40
1000 cells/millimeters cubed (mm^3)
  ANC | 1.2 [0 to 5]
  Platelets | 78 [6 to 184]
  WBC count | 2.3 [1 to 6]

17. Secondary Outcome: Nadir Values for Hemoglobin, a Hematologic Parameter
Description: Nadir is defined as the lowest laboratory value recorded following the administration of study medication. Hemoglobin is the iron-containing oxygen-transport metalloprotein in the red blood cells.
Time Frame: as for outcome 1
Population: as for outcome 16
Measure: Median (Full Range); unit: g/dL
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 40
g/dL | 11.3 [7 to 15]

18. Secondary Outcome: Number of Participants Who Became Positive or Negative for Human Anti-murine Antibody (HAMA) After Study Treatment
Description: Tositumomab is a murine (mouse) antibody. Participants in this study were evaluated to determine if they developed a human anti-murine antibody (HAMA) immune response after administration of tositumomab and iodine I 131 tositumomab.
Time Frame: as for outcome 1
Population: ITT Exposed Population
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 41
participants
  Positive | 4
  Negative | 37

19. Secondary Outcome: Time to HAMA Positivity From First Dosimetric Dose
Description: Time to HAMA positivity is defined as the time from the first dosimetric dose to the first reported HAMA-positive result for the participant.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Participants who converted to HAMA positivity were analyzed.
Measure: Median (Full Range); unit: days
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 4
days | 112 [12 to 264]

20. Secondary Outcome: Number of Participants in the Indicated Categories of Thyroid Function Assessment
Description: Hypothyroidism, a condition in which the thyroid gland does not produce enough thyroid hormone (resulting in the elevation of thyroid stimulating hormone [TSH] in the blood), may result from treatment with radioactive iodine I 131. A thyroid blockade medication was given prior to administration of the study drug and up to 2 weeks after the therapeutic dose to prevent the uptake of I 131 in the thyroid gland. Thyroid function was determined periodically, including during follow-up, in order to assess if there was any effect of the I 131 on thyroid function, such as hypothyroidism.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Participants who were evaluable for thyroid function assessment and who had no elevated TSH level or hypothyroidism at baseline were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 36
participants
  Elevated TSH post therapy | 9
  Hypothyroidism | 3

21. Secondary Outcome: Number of Days Each Participant Took to Reach Hypothyroidism After the First Dosimetric Dose
Description: Hypothyroidism is a condition in which the thyroid gland does not produce enough thyroid hormone (resulting in the elevation of thyroid stimulating hormone [TSH] in the blood).
Time Frame: as for outcome 1
Population: ITT Exposed Population. Participants experiencing hypothyroidism were analyzed.
Measure: Number; unit: days
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 3
days
  Participant Number 19/73 | 192
  Participant Number 18/68 | 475
  Participant Number 19/57 | 671

ADVERSE EVENTS:
Time Frame: Par. were evaluated until death/disease progression or 2 years in Study BEX104505. Par. who completed 2 years in BEX104505 were followed in study BEX104528 for up to 125 months. Data are included from both Study BEX104505 and Study BEX104528.
Arm/Group | TST and Iodine I 131 TST
Serious Adverse Events (participants affected / at risk) | 13/41
Other Adverse Events (participants affected / at risk) | 40/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TST and Iodine I 131 TST (N=41)
Anemia (Blood and lymphatic system disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Pancytopenia (Blood and lymphatic system disorders) | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Lower Respiratory Tract Infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Hemophilus Infection (Infections and infestations) | 1
Herpes Simplex (Infections and infestations) | 1
Herpes Zoster (Infections and infestations) | 1
Neutropenic Sepsis (Infections and infestations) | 1
Respiratory Tract Infection (Infections and infestations) | 1
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Pyrexia (General disorders) | 2
Hematuria (Renal and urinary disorders) | 1
Renal Failure Chronic (Renal and urinary disorders) | 1
Hepatic Failure (Hepatobiliary disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Radiculitis Brachial (Nervous system disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TST and Iodine I 131 TST (N=41)
Nausea (Gastrointestinal disorders) | 13
Constipation (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 3
Abdominal Discomfort (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 1
Aphthous Stomatitis (Gastrointestinal disorders) | 1
Cheilosis (Gastrointestinal disorders) | 1
Epigastric Discomfort (Gastrointestinal disorders) | 1
Gastrointestinal Disorder (Gastrointestinal disorders) | 1
Gingival Bleeding (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Tongue Coated (Gastrointestinal disorders) | 1
ANC <1000 cells/cubic millimeters (10^3/mm^3) (Investigations) | 18
Platelets <50000 cells/10^3/mm^3 (Investigations) | 15
WBC <2000 cells/10^3/mm^3 (Investigations) | 14
Hemoglobin <8.0 g/dL (Investigations) | 3
Fatigue (General disorders) | 8
Chills (General disorders) | 5
Pyrexia (General disorders) | 5
Edema Peripheral (General disorders) | 4
Pain (General disorders) | 4
Chest Discomfort (General disorders) | 2
Chest Pain (General disorders) | 2
Asthenia (General disorders) | 1
Feeling Cold (General disorders) | 1
Gait Disturbance (General disorders) | 1
Ill-defined Disorder (General disorders) | 1
Influenza Like Illness (General disorders) | 1
Local Swelling (General disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 5
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 6
Herpes Zoster (Infections and infestations) | 2
Lower Respiratory Tract Infection (Infections and infestations) | 2
Respiratory Tract Infection (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Herpes Simplex (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Infusion Site Infection (Infections and infestations) | 1
Neutropenic Sepsis (Infections and infestations) | 1
Oral Herpes (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Viral Infection (Infections and infestations) | 1
Headache (Nervous system disorders) | 7
Lethargy (Nervous system disorders) | 7
Paraesthesia (Nervous system disorders) | 3
Somnolence (Nervous system disorders) | 3
Ageusia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dizziness Postural (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Post Herpetic Neuralgia (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Productive Cough (Reproductive system and breast disorders) | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 4
Erythema (Skin and subcutaneous tissue disorders) | 2
Petechiae (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Subcutaneous Nodule (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Anemia (Blood and lymphatic system disorders) | 1
Lymph Node Pain (Blood and lymphatic system disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 2
Muscle Injury (Injury, poisoning and procedural complications) | 1
Skeletal Injury (Injury, poisoning and procedural complications) | 1
Hypothyroidism (Endocrine disorders) | 5
Orthostatic Hypotension (Vascular disorders) | 2
Flushing (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 3
Dysuria (Renal and urinary disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Palpitations (Cardiac disorders) | 2
Conjunctival Hemorrhage (Eye disorders) | 1
Dry Eye (Eye disorders) | 1
Insomnia (Psychiatric disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Hypersensitivity (Immune system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.